CLINICAL TRIAL: NCT00003015
Title: Ultimate Low Grade Glioma Study
Brief Title: Carboplatin Plus Vincristine in Treating Children and Adolescents With Low Grade Glioma
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Societe Internationale d'Oncologie Pediatrique (Other)
Organization: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: CDR0000065595; SIOP-95-2; EU-96063
Record Dates: First submitted 1999-11-01; First posted 2004-05-27 (Estimated); Last update posted 2013-12-04 (Estimated); Status verified 2001-01

CONDITIONS: Brain and Central Nervous System Tumors
Keywords: childhood low-grade cerebral astrocytoma; childhood oligodendroglioma; untreated childhood visual pathway glioma; untreated childhood cerebellar astrocytoma
MeSH Terms: conditions — Central Nervous System Neoplasms; Oligodendroglioma | interventions — Carboplatin; Vincristine; Radiotherapy

INTERVENTIONS:
Drug: carboplatin
Drug: vincristine sulfate
Procedure: conventional surgery
Radiation: radiation therapy

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Combining more than one drug may kill more tumor cells.

PURPOSE: Randomized phase III trial to compare the effectiveness of carboplatin plus vincristine in treating children and adolescents with low grade glioma.

DETAILED DESCRIPTION:
OBJECTIVES: I. Develop a standardized scheme of therapy for children and adolescents with low grade glioma. II. Determine the effectiveness of carboplatin and vincristine in treating children aged less than 5 years with severe or progressive symptoms or unequivocal imaging evidence of tumor growth.

OUTLINE: A complete resection of tumor is performed on patients with low grade glioma with or without neurofibromatosis type 1. Surgery is reconsidered following tumor relapse, progression, or clinical deterioration. Every effort is made to obtain a biopsy from patients not receiving debulking surgery. Nonoperative patients and postoperative patients who are not candidates for second surgery receive chemotherapy or radiotherapy. Postoperative patients receive radiotherapy following surgical wound healing and within 28 days of resection. Children less than 5 years old receive chemotherapy first, then radiotherapy if the tumor subsequently progresses or recurs. All other patients receive radiotherapy, then chemotherapy. The latter treatment is conducted in the presence of tumor progression. Chemotherapy is given in 2 parts, first an initial intensive phase (phase 1), then a later continuation phase (phase 2). In phase 1, patients receive vincristine IV weekly for 10 weeks and carboplatin IV every 3 weeks. In phase 2, patients receive vincristine IV and carboplatin IV every 4 weeks for a total treatment time of 52 weeks. Chemotherapy continues until disease progression or unacceptable toxicity. Patients receive radiotherapy daily 5 times a week. Patients are followed every 3 months for 1 year, every 6 months for 1 year, and then annually for 3 years.

PROJECTED ACCRUAL: A total of 200 patients will be accrued for this study over 5 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Patients with or without neurofibromatosis type 1 (NF1) with low grade glioma not previously treated with chemotherapy or radiotherapy Tumor types considered are: Low grade astrocytoma (Kernohan grade 1/2) Oligodendroglioma Mixed oligoastrocytoma Ganglioglioma Patients with NF1 and hypothalamic/visual pathway glioma are eligible without biopsy All CNS sites are eligible, including biopsy proven low grade spinal tumors and intrinsic brain stem tumors No malignant (anaplastic) glioma (Kernohan grade 3/4), glioblastoma multiforme, and ependymal tumors

PATIENT CHARACTERISTICS: Age: Under 16 Performance status: Not specified Life expectancy: Not specified Hematopoietic: Not specified Hepatic: Not specified Renal: Not specified

PRIOR CONCURRENT THERAPY: Biologic therapy: Not specified Chemotherapy: See Disease Characteristics Endocrine therapy: Not specified Radiotherapy: See Disease Characteristics Surgery: Not specified

Max Age: 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 200 (Estimated)
Dates: Start 1997-01

CONTACTS AND LOCATIONS:
Overall Officials: David A. Walker, Study Chair — Queen's Medical Center
Locations (3):
- Zentralklinikum Augsburg, Augsburg, Germany
- University of Padua, Padua, Italy
- Queen's Medical Centre, Nottingham, England, United Kingdom

REFERENCES:
- [Result] Gnekow AK, Perilongo G, Zanetti I, et al.: Single dose carboplatin and vincristine (VER) for progressive low-grade glioma (LGG) in childhood. A SIOP/GPOH study. [Abstract] International Symposium on Pediatric Neuro-Oncology, May 18-21, 1994, Houston, Tx. A-89, 1999.